CLINICAL TRIAL: NCT01096862
Title: A Phase 2a, Randomized, Double-blind, Placebo-Controlled, Sequential Group, Multiple-Dose Escalation Study to Evaluate the Efficacy and Safety of ASP015K in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Explore Efficacy and Safety of ASP015K in Subjects With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 015K-CL-PS01
Record Dates: First submitted 2010-03-18; First posted 2010-03-31 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Psoriasis
Keywords: ASP015K; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — peficitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): lowest dose
  Interventions: Drug: peficitinib
- Group 2 (Experimental): low dose
  Interventions: Drug: peficitinib
- Group 3 (Experimental): high dose
  Interventions: Drug: peficitinib
- Group 4 (Experimental): highest dose
  Interventions: Drug: peficitinib
- Group 5 (Experimental): medium dose
  Interventions: Drug: peficitinib
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: peficitinib — oral
  Other Names: ASP015K
  Arms: Group 1; Group 2; Group 3; Group 4; Group 5
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to explore the efficacy and safety of multiple, escalating doses of ASP015K when compared to placebo in subjects with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
Following completion of at least 1 week of study drug for all subjects in group 1, the Sponsor will review the safety information of these subjects prior to enrolling off-treatment subjects into the next dose group. Dose escalation will continue in this manner (unless stopping criteria are met) until all groups have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has moderate to severe plaque psoriasis for 6 months or longer with at least 10% Body Surface Area (BSA) affected
* Subject must be a candidate for phototherapy and/or systemic therapy

Exclusion Criteria:

* Subject has non-plaque psoriasis or drug-induced psoriasis
* Subject is on systemic psoriasis therapy within 56 days or 5 half-lives, whichever is longer, prior to first dose of study drug
* Subject has a positive TB skin test within 3 months of screening or at screening
* Subject has an abnormal chest x-ray

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2010-03-23 (Actual); Primary Completion 2011-07-27 (Actual); Study Completion 2011-07-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the end of treatment in Psoriasis Area Severity Index (PASI) score | 6 weeks
Safety assessed from baseline to end of treatment by recording adverse events, physical examinations, vital signs, laboratory assessments and electrocardiograms (ECGs) | 6 weeks

SECONDARY OUTCOMES:
Change from baseline to end of treatment in Physicians Static Global Assessment (PSGA) | 6 weeks
Change from baseline to end of treatment in percent body surface area (BSA) | 6 weeks
Success of the treatment of psoriasis as measured by a Physician's Static Global Assessment (PSGA) of Almost Clear or Clear | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (11):
- United States (11):
  - Total Skin & Beauty Dermatology Center, Birmingham, Alabama
  - Therapeutics Clinical Research, San Diego, California
  - FXM Research, Corp., Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Derm Research, PLLC, Louisville, Kentucky
  - Oregon Medical Research Center, Portland, Oregon
  - Palmetto Clinical Trial Services, Greenville, South Carolina
  - Rivergate Dermatology, Goodlettsville, Tennessee
  - J & S Studies, College Station, Texas
  - Virginia Clinical Research, Norfolk, Virginia
  - Madison Skin & Research, Inc, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Papp K, Pariser D, Catlin M, Wierz G, Ball G, Akinlade B, Zeiher B, Krueger JG. A phase 2a randomized, double-blind, placebo-controlled, sequential dose-escalation study to evaluate the efficacy and safety of ASP015K, a novel Janus kinase inhibitor, in patients with moderate-to-severe psoriasis. Br J Dermatol. 2015 Sep;173(3):767-76. doi: 10.1111/bjd.13745. Epub 2015 Jun 19. PMID 25704750
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=327